CLINICAL TRIAL: NCT07037303
Title: Comparison of Effectiveness Between Active Cycle of Breathing Techniques (ACBT) and Oscillating Positive Expiratory Pressure (OPEP, Aerobika) Device Assisted Treatment in Patients With Bronchiectasis in Korea : Randomized Controlled Trials
Brief Title: Comparing Active Cycle of Breathing Techniques (ACBT) and Aerobika in Treating Bronchiectasis in Korea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chungbuk National University Hospital (Other)
Collaborators: Trudell Medical International (Industry)
Responsible Party: Principal Investigator, Bumhee Yang, MD, Associate professor, Chungbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB No. 2025-02-031
Record Dates: First submitted 2025-06-03; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Bronchiectasis; Bronchiectasis With Acute Exacerbation
Keywords: bronchiectasis; aerobika; ACBT
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Cycle of Breathing Technique (ACBT) group (Active Comparator): patients with bronchiectasis using ACBT
  Interventions: Device: Active Cycle of Breathing Technique (ACBT) group
- Active Cycle of Breathing Technique (ACBT) and Oscillatory Positive Expiratory Pressure (OPEP) group (Experimental): Patients with bronchiectasis using ACBT and OPEP simultaneously
  Interventions: Device: Active Cycle of Breathing Technique (ACBT) and Oscillatory Positive Expiratory Pressure (OPEP) group

INTERVENTIONS:
Device: Active Cycle of Breathing Technique (ACBT) and Oscillatory Positive Expiratory Pressure (OPEP) group — Patients with bronchiectasis using ACT and OPEP simultaneously
  Arms: Active Cycle of Breathing Technique (ACBT) and Oscillatory Positive Expiratory Pressure (OPEP) group
Device: Active Cycle of Breathing Technique (ACBT) group — Patients will receive only ACBT for airway clearance.
  Arms: Active Cycle of Breathing Technique (ACBT) group

SUMMARY:
Title:

Comparison of Effectiveness Between Active Cycle of Breathing Techniques (ACBT) and Oscillating Positive Expiratory Pressure (OPEP, Aerobika) Device Assisted Treatment in Patients With Bronchiectasis in Korea: A Randomized Controlled Trial

Purpose:

This study aims to evaluate the effectiveness of Active Cycle of Breathing Techniques (ACBT) alone versus ACBT combined with an Oscillating Positive Expiratory Pressure (OPEP) device (Aerobika) in patients with bronchiectasis. The goal is to determine whether the combination therapy reduces the frequency of acute exacerbations and improves patient symptoms compared to ACBT alone.

Primary Questions:

Does the use of ACBT plus Aerobika reduce the number of acute exacerbations in patients with bronchiectasis who experience ≥3 exacerbations per year?

What symptoms and adverse events are observed in participants using the Aerobika device?

Study Design:

This is a single-center, randomized, controlled clinical trial conducted at Chungbuk National University Hospital in Korea. 100 adult patients diagnosed with bronchiectasis and having ≥3 acute exacerbations within 1 year will be enrolled and randomized into two groups (1:1):

Active Cycle of Breathing Technique (ACBT) group

Active Cycle of Breathing Technique (ACBT) and Oscillatory Positive Expiratory Pressure (OPEP) group

The intervention period lasts 12 months, with clinic visits scheduled at 0, 1, 3, 6, 9, and 12 months.

Participation Involves:

Use of ACBT with or without Aerobika daily for 12 months

In-person clinic visits every 1 to 3 months

Monthly phone follow-ups to assess symptoms and adverse events

Completion of questionnaires (mMRC, BHQ, CAT) and clinical tests including PFT and laboratory tests

Tracking of exacerbation frequency, sputum volume, and quality

DETAILED DESCRIPTION:
Primary Questions:

Does the use of ACBT plus Aerobika reduce the number of acute exacerbations in patients with bronchiectasis who experience ≥3 exacerbations per year?

Answer) To date, no studies have demonstrated that the use of ACBT plus Aerobika reduces acute exacerbations in patients with bronchiectasis who experience frequent exacerbations.

What symptoms and adverse events are observed in participants using the Aerobika device?

Answer) Oscillating PEP devices are not recommended in patients with neuromuscular weakness, recent head and neck surgery or trauma, active hemoptysis, untreated pneumothorax, and middle ear disease

Ref. Coppolo DP, Schloss J, Suggett JA, Mitchell JP. Non-Pharmaceutical Techniques for Obstructive Airway Clearance Focusing on the Role of Oscillating Positive Expiratory Pressure (OPEP): A Narrative Review. Pulm Ther. (2022) 8:1-41.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients diagnosed with bronchiectasis involving one or more lobes on chest computed tomography (CT)
* Patients experiencing frequent exacerbations (3 or more exacerbations) within 1 year
* Patients able and willing to use the Aerobika device (OPEP)

Exclusion Criteria:

* Diagnosis of bronchiectasis due to cystic fibrosis
* Traction bronchiectasis due to interstitial lung disease (ILD)
* Pregnant patients
* Patients with a history of OPEP device use
* Patients who cannot tolerate increased breathing work
* Hemodynamic instability (e.g., unstable blood pressure)
* Patients with a past or current history of hemoptysis (pulmonary bleeding) and untreated pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Acute Exacerbations in Patients with Bronchiectasis | 12 months from baseline
  Number of acute exacerbations experienced by patients diagnosed with bronchiectasis during the 12-month study period.

SECONDARY OUTCOMES:
Improvement in subjective symptoms (1) | Subjective symptoms: 1, 3, 6, 9, and 12 months from baseline
  Evaluation of reductions from baseline in patients' self-reported symptoms (using Modified Medical Research Council (mMRC) dyspnea scale score) assessed at 1, 3, 6, 9, and 12 months (range: 0-4; higher scores indicate worse dyspnea)
Improvement in subjective symptoms (2) | Subjective symptoms: 1, 3, 6, 9, and 12 months from baseline
  Evaluation of changes from baseline in patients' self-reported symptoms (using Bronchiectasis Health Questionnaire (BHQ) score) assessed at 1, 3, 6, 9, and 12 months (range: 0-100; higher scores indicate better health status or quality of life)
Improvement in subjective symptoms (3) | Subjective symptoms: 1, 3, 6, 9, and 12 months from baseline
  Evaluation of reductions from baseline in patients' self-reported symptoms (using COPD Assessment Test (CAT) score) assessed at 1, 3, 6, 9, and 12 months (range: 0-40; higher scores indicate worse health status or greater impact of COPD symptoms)
Improvement in objective assessment | Forced Vital Capacity (FVC) measured in liters (L): 12 months from baseline
  Evaluation of changes from baseline in patients' pulmonary function, specifically Forced Vital Capacity (FVC) measured in liters (L), at 12 months.
Improvement in objective assessment | Forced Vital Capacity (FVC) expressed as a percentage of predicted value (FVC %): 12 months from baseline
  Evaluation of changes from baseline in patients' pulmonary function, specifically Forced Vital Capacity (FVC) expressed as a percentage of predicted value (FVC %), measured at 12 months.
Improvement in objective assessment | Forced Expiratory Volume in 1 second (FEV1) measured in liters (L): 12 months from baseline
  Evaluation of changes from baseline in patients' pulmonary function, specifically Forced Expiratory Volume in 1 second (FEV1) measured in liters (L), at 12 months.
Improvement in objective assessment | Forced Expiratory Volume in 1 second (FEV1) expressed as a percentage of predicted value (FEV1 %): 12 months from baseline
  Evaluation of changes from baseline in patients' pulmonary function, specifically Forced Expiratory Volume in 1 second (FEV1) expressed as a percentage of predicted value (FEV1 %), measured at 12 months.
Improvement in objective assessment | the ratio of Forced Expiratory Volume in 1 second to Forced Vital Capacity (FEV1/FVC): 12 months from baseline
  Evaluation of changes from baseline in patients' pulmonary function, specifically the ratio of Forced Expiratory Volume in 1 second to Forced Vital Capacity (FEV1/FVC), measured at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SR, Kim SH, Kim GH, Cho JY, Choi H, Lee H, Ra SW, Lee KM, Choe KH, Oh YM, Shin YM, Yang B. Effectiveness of the use of an oscillating positive expiratory pressure device in bronchiectasis with frequent exacerbations: a single-arm pilot study. Front Med (Lausanne). 2023 May 12;10:1159227. doi: 10.3389/fmed.2023.1159227. eCollection 2023. PMID 37250647
- [Background] Yang B, Choi H, Lim JH, Park HY, Kang D, Cho J, Lee JS, Lee SW, Oh YM, Moon JY, Kim SH, Kim TH, Sohn JW, Yoon HJ, Lee H. The disease burden of bronchiectasis in comparison with chronic obstructive pulmonary disease: a national database study in Korea. Ann Transl Med. 2019 Dec;7(23):770. doi: 10.21037/atm.2019.11.55. PMID 32042786
- [Background] Chalmers JD, Chang AB, Chotirmall SH, Dhar R, McShane PJ. Bronchiectasis. Nat Rev Dis Primers. 2018 Nov 15;4(1):45. doi: 10.1038/s41572-018-0042-3. PMID 30442957
- [Background] Hill AT, Sullivan AL, Chalmers JD, De Soyza A, Elborn SJ, Floto AR, Grillo L, Gruffydd-Jones K, Harvey A, Haworth CS, Hiscocks E, Hurst JR, Johnson C, Kelleher PW, Bedi P, Payne K, Saleh H, Screaton NJ, Smith M, Tunney M, Whitters D, Wilson R, Loebinger MR. British Thoracic Society Guideline for bronchiectasis in adults. Thorax. 2019 Jan;74(Suppl 1):1-69. doi: 10.1136/thoraxjnl-2018-212463. No abstract available. PMID 30545985

DOCUMENTS (1):
  • Study Protocol (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT07037303/Prot_000.pdf